CLINICAL TRIAL: NCT02683447
Title: Impact of Acute Care Physician's Age on Crisis Management Performance and Learning After Simulation-based Education
Brief Title: Ageing and Acute Care Physicians' Performance
Status: Completed | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: University of Toronto (Other); University of Ottawa (Other)
Responsible Party: Principal Investigator, Dr. Fahad Alam, Anesthesiologist, Sunnybrook Health Sciences Centre
Other Study IDs: 140-2015
Record Dates: First submitted 2016-02-09; First posted 2016-02-17 (Estimated); Results first posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2024-12

CONDITIONS: Ageing
Keywords: Continuing Medical Education; Simulation; Non-technical Skills; Crisis Resource Management

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CRM Simulation: Each participant will manage a PEA arrest scenario (pre-test) and then be debriefed on their CRM skills by a trained facilitator for 20 minutes. They will then manage another crisis scenario (PEA arrest with a different inciting event) as an immediate post-test. Three months afterwards participants will return to manage a third PEA arrest scenario, which will serve as a retention post-test.
  Interventions: Other: CRM Simulation

INTERVENTIONS:
Other: CRM Simulation — Each participant will manage a PEA arrest scenario (pre-test) and then be debriefed on their CRM skills by a trained facilitator for 20 minutes. They will then manage another crisis scenario (PEA arrest with a different inciting event) as an immediate post-test. Three months afterwards participants will return to manage a third PEA arrest scenario, which will serve as a retention post-test.

SUMMARY:
The proportion of older acute care physicians (ACPs) has been increasing. Ageing is associated with physiological changes and research investigating how such age-related physiological changes affect clinical performance is lacking. Specifically, Crisis Resource Management (CRM) consists of essential clinical skills in acute care specialties which when absent, can significantly impact patient safety. As such, the goals of this study are to investigate whether ageing has a correlation with baseline CRM skills of ACPs and whether ageing influences learning from high fidelity simulation.

DETAILED DESCRIPTION:
The proportion of older acute care physicians (ACP), emergency, critical care & anesthesia, has been steadily increasing. Ageing is associated with physiological changes, which in turn can influence a physician's clinical abilities and decision-making. The litigation and physician disciplinary data suggests that incidents involving all physicians are likely to occur later in practice, with degree of injury identified in the claims being of greater severity. However research, investigating how age-related physiological changes affect clinical performance and patient safety, is lacking.

CRM skills are essential skills within acute care specialties, and are vital for patient safety. CRM encompasses technical skills, as well as a rapid and organized approach to non-technical, cognitive skills such as decision-making, task management, situational awareness and team management. High-fidelity full body mannequin simulation-based education is effective for learning CRM, including transfer of skills from the simulated setting to the clinical setting and improving patient outcome. However, there is a gap in the literature on whether physicians' age influences baseline CRM performance and also learning from simulation-based education.

Although the effectiveness of high-fidelity simulation-based education has been studied extensively in junior learner populations (students, residents, fellows), there are a limited number of studies investigating its effectiveness in teaching CRM in the ageing physician population. In fact, a recent systematic review looking at the role of simulation in continuing medical education (CME) in ACPs supported that there is limited evidence supporting improved learning. Despite not knowing whether simulation is the correct tool in an ageing population, it is being recommended as a training, regulation and assessment tool for practicing physicians.

Objectives:

The goals of this study are to:

1. Investigate whether ageing has a correlation with baseline CRM skills of ACPs using simulated crisis scenarios and
2. Assess whether ageing influences learning from high fidelity simulation.

ELIGIBILITY:
Inclusion Criteria:

* Emergency physicians
* Critical care physicians
* Anesthesiologists
* minimum 5 years of practice post-residency

Exclusion Criteria:

* Post-call day of participation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Practicing emergency, critical care and anesthesia staff with a minimum 5 years of practice post residency will be approached for participation.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fahad Alam, MD, FRCPC, Principal Investigator — Sunnybrook Health Sciences Centre; Sylvain Boet, MD, MEd, PhD, Principal Investigator — University of Ottawa
Locations (2):
- Canada (2):
  - University of Ottawa, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Katz JD. Issues of concern for the aging anesthesiologist. Anesth Analg. 2001 Jun;92(6):1487-92. doi: 10.1097/00000539-200106000-00027. No abstract available. PMID 11375831
- [Background] Baxter AD, Boet S, Reid D, Skidmore G. The aging anesthesiologist: a narrative review and suggested strategies. Can J Anaesth. 2014 Sep;61(9):865-75. doi: 10.1007/s12630-014-0194-x. Epub 2014 Jul 2. PMID 24985937
- [Background] Baird M, Daugherty L, Kumar KB, Arifkhanova A. Regional and Gender Differences and Trends in the Anesthesiologist Workforce. Anesthesiology. 2015 Nov;123(5):997-1012. doi: 10.1097/ALN.0000000000000834. PMID 26291778
- [Background] Siu LW, Boet S, Borges BC, Bruppacher HR, LeBlanc V, Naik VN, Riem N, Chandra DB, Joo HS. High-fidelity simulation demonstrates the influence of anesthesiologists' age and years from residency on emergency cricothyroidotomy skills. Anesth Analg. 2010 Oct;111(4):955-60. doi: 10.1213/ANE.0b013e3181ee7f4f. Epub 2010 Aug 24. PMID 20736429
- [Background] Daugherty L, Fonseca R, Kumar KB, Michaud PC. An Analysis of the Labor Markets for Anesthesiology. Rand Health Q. 2011 Sep 1;1(3):18. eCollection 2011 Fall. PMID 28083205
- [Background] Duke, E. (2006). The Critical Care Workforce: A Study of the Supply and Demand for Critical Care Physicians : Report to Congress (p. 36). U.S. Department of Health & Human Sciences.
- [Background] Durning SJ, Artino AR, Holmboe E, Beckman TJ, van der Vleuten C, Schuwirth L. Aging and cognitive performance: challenges and implications for physicians practicing in the 21st century. J Contin Educ Health Prof. 2010 Summer;30(3):153-60. doi: 10.1002/chp.20075. PMID 20872769
- [Background] Eva KW. The aging physician: changes in cognitive processing and their impact on medical practice. Acad Med. 2002 Oct;77(10 Suppl):S1-6. doi: 10.1097/00001888-200210001-00002. No abstract available. PMID 12377689
- [Background] Trunkey DD, Botney R. Assessing competency: a tale of two professions. J Am Coll Surg. 2001 Mar;192(3):385-95. doi: 10.1016/s1072-7515(01)00770-0. No abstract available. PMID 11245381
- [Background] Turnbull J, Carbotte R, Hanna E, Norman G, Cunnington J, Ferguson B, Kaigas T. Cognitive difficulty in physicians. Acad Med. 2000 Feb;75(2):177-81. doi: 10.1097/00001888-200002000-00018. PMID 10693852
- [Background] Norman G, Young M, Brooks L. Non-analytical models of clinical reasoning: the role of experience. Med Educ. 2007 Dec;41(12):1140-5. doi: 10.1111/j.1365-2923.2007.02914.x. Epub 2007 Nov 13. PMID 18004990
- [Background] Tessler MJ, Shrier I, Steele RJ. Association between anesthesiologist age and litigation. Anesthesiology. 2012 Mar;116(3):574-9. doi: 10.1097/ALN.0b013e3182475ebf. PMID 22354239
- [Background] Alam A, Khan J, Liu J, Klemensberg J, Griesman J, Bell CM. Characteristics and rates of disciplinary findings amongst anesthesiologists by professional colleges in Canada. Can J Anaesth. 2013 Oct;60(10):1013-9. doi: 10.1007/s12630-013-0006-8. Epub 2013 Jul 30. PMID 23897490
- [Background] Duclos A, Peix JL, Colin C, Kraimps JL, Menegaux F, Pattou F, Sebag F, Touzet S, Bourdy S, Voirin N, Lifante JC; CATHY Study Group. Influence of experience on performance of individual surgeons in thyroid surgery: prospective cross sectional multicentre study. BMJ. 2012 Jan 10;344:d8041. doi: 10.1136/bmj.d8041. PMID 22236412
- [Background] Khaliq AA, Dimassi H, Huang CY, Narine L, Smego RA Jr. Disciplinary action against physicians: who is likely to get disciplined? Am J Med. 2005 Jul;118(7):773-7. doi: 10.1016/j.amjmed.2005.01.051. PMID 15989912
- [Background] Boet S, Bould MD, Fung L, Qosa H, Perrier L, Tavares W, Reeves S, Tricco AC. Transfer of learning and patient outcome in simulated crisis resource management: a systematic review. Can J Anaesth. 2014 Jun;61(6):571-82. doi: 10.1007/s12630-014-0143-8. Epub 2014 Mar 25. PMID 24664414
- [Background] Marinopoulos SS, Dorman T, Ratanawongsa N, Wilson LM, Ashar BH, Magaziner JL, Miller RG, Thomas PA, Prokopowicz GP, Qayyum R, Bass EB. Effectiveness of continuing medical education. Evid Rep Technol Assess (Full Rep). 2007 Jan;(149):1-69. PMID 17764217
- [Background] Khanduja PK, Bould MD, Naik VN, Hladkowicz E, Boet S. The role of simulation in continuing medical education for acute care physicians: a systematic review. Crit Care Med. 2015 Jan;43(1):186-93. doi: 10.1097/CCM.0000000000000672. PMID 25343571
- [Background] Steadman RH. Improving on reality: can simulation facilitate practice change? Anesthesiology. 2010 Apr;112(4):775-6. doi: 10.1097/ALN.0b013e3181d3e337. No abstract available. PMID 20216388
- [Background] Curtis MT, DiazGranados D, Feldman M. Judicious use of simulation technology in continuing medical education. J Contin Educ Health Prof. 2012 Fall;32(4):255-60. doi: 10.1002/chp.21153. PMID 23280528
- [Background] Savoldelli GL, Naik VN, Hamstra SJ, Morgan PJ. Barriers to use of simulation-based education. Can J Anaesth. 2005 Nov;52(9):944-50. doi: 10.1007/BF03022056. PMID 16251560
- [Background] Davis DA, Mazmanian PE, Fordis M, Van Harrison R, Thorpe KE, Perrier L. Accuracy of physician self-assessment compared with observed measures of competence: a systematic review. JAMA. 2006 Sep 6;296(9):1094-102. doi: 10.1001/jama.296.9.1094. PMID 16954489
- [Background] Kim J, Neilipovitz D, Cardinal P, Chiu M, Clinch J. A pilot study using high-fidelity simulation to formally evaluate performance in the resuscitation of critically ill patients: The University of Ottawa Critical Care Medicine, High-Fidelity Simulation, and Crisis Resource Management I Study. Crit Care Med. 2006 Aug;34(8):2167-74. doi: 10.1097/01.CCM.0000229877.45125.CC. PMID 16775567
- [Background] McEvoy MD, Smalley JC, Nietert PJ, Field LC, Furse CM, Blenko JW, Cobb BG, Walters JL, Pendarvis A, Dalal NS, Schaefer JJ 3rd. Validation of a detailed scoring checklist for use during advanced cardiac life support certification. Simul Healthc. 2012 Aug;7(4):222-35. doi: 10.1097/SIH.0b013e3182590b07. PMID 22863996
- [Derived] Alam F, LeBlanc VR, Baxter A, Tarshis J, Piquette D, Gu Y, Filipowska C, Krywenky A, Kester-Greene N, Cardinal P, Au S, Lam S, Boet S, Clinical Trials Group PA. Does the age of acute care physicians impact their (1) crisis management performance and (2) learning after simulation-based education? A protocol for a multicentre prospective cohort study in Toronto and Ottawa, Canada. BMJ Open. 2018 Apr 21;8(4):e020940. doi: 10.1136/bmjopen-2017-020940. PMID 29680811

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CRM Simulation
Started | 48
Completed | 46
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | CRM Simulation
Number analyzed (Participants) | 48
Age, Continuous [Mean (Full Range); unit: years] | 49.5 [34.0 to 71.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Age, Categorical [Count of Participants; unit: Participants]
  <45 | 15
  45-54 | 20
  55-64 | 10
  65+ | 3
Biological Age, Continuous [Mean (Full Range); unit: years] — Participants completed a questionnaire to determine their biological age (www.projectbiglife.ca)
  years | 43.4 [27.4 to 66.5]
Biological Age, Categorical [Count of Participants; unit: Participants]
  <45 | 32
  45-54 | 9
  55-64 | 4
  65+ | 3
Enrollment Site [Count of Participants; unit: Participants]
  University of Toronto | 34
  University of Ottawa | 14
Specialty [Count of Participants; unit: Participants]
  Anesthesia | 35
  Emergency | 8
  Intensive care | 5
Years in Practice [Count of Participants; unit: Participants]
  0-10 | 10
  11-20 | 20
  21-30 | 13
  31-40 | 4
  41-50 | 0
  >50 | 1
Previous Full-body Manikin Simulation Scenarios Completed [Count of Participants; unit: Participants]
  0-5 | 28
  6-10 | 9
  11-15 | 7
  16-20 | 0
  >20 | 4
What Percentage of Practice Time do you Manage ACLS Crises? [Count of Participants; unit: Participants]
  0-10% | 36
  11-20% | 9
  21-30% | 0
  31-40% | 1
  41-50% | 0
  >50% | 2
Have you ever been an ACLS Instructor? [Count of Participants; unit: Participants]
  Yes | 10
  No | 38

OUTCOME MEASURES:

1. Primary Outcome: CRM Performance During First Sim Scenario Assessed by Ottawa Global Rating Scale (GRS)
Description: Ottawa GRS score correlated with chronological age. The Ottawa GRS assesses non-technical CRM skills on a 7-point scale (minimum 1, maximum 7), with higher scores indicating better performance.
Time Frame: After managing first simulation scenario - Day 1
Measure: Number; unit: Pearson correlation coefficient
Arm/Group | CRM Simulation
Number analyzed (Participants) | 48
Pearson correlation coefficient | -0.299
Statistical Analysis 1: Comparison: CRM Simulation; Test type: Other — Correlation; p = 0.039, Pearson correlation — P < 0.05 is considered statistically significant

2. Primary Outcome: CRM Performance During First Sim Scenario Assessed by ACLS Checklist
Description: ACLS (Advanced Cardiac Life Support) score will be correlated with chronological age. Items on the checklist were separated into two components: 1) the ACLS correct score (minimum score 0, maximum score 30), where higher scores indicate better performance, and 2) the ACLS risk score (minimum score 0, maximum score 17) where higher scores indicate worse performance.
Time Frame: After managing first simulation scenario - Day 1
Measure: Number; unit: Pearson correlation coefficient
Arm/Group | CRM Simulation
Number analyzed (Participants) | 48
Pearson correlation coefficient
  ACLS correct score | -0.438
  ACLS risk score | 0.143
Statistical Analysis 1: Comparison: CRM Simulation; ACLS correct score; Test type: Other — Correlation; p < 0.01, Pearson correlation — P < 0.05 is considered statically significant
Statistical Analysis 2: Comparison: CRM Simulation; ACLS risk score; Test type: Other — Correlation; p = 0.322, Pearson correlation — P < 0.05 is considered statically significant

3. Secondary Outcome: Learning From High-fidelity Simulation Education Assessed by Ottawa Global Rating Scale
Description: Ottawa GRS score will be compared to score in first scenario to look for improvement. The Ottawa GRS assesses non-technical CRM skills on a 7-point scale (minimum 1, maximum 7), with higher scores indicating better performance. The mean difference in GRS score between pre-test (scenario 1) and immediate post-test (scenario 2) is reported.
Time Frame: After managing second simulation scenario - Day 1
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | CRM Simulation
Number analyzed (Participants) | 48
Score on a scale | 2.28 [1.14 to 3.42]

4. Secondary Outcome: Learning From High-fidelity Simulation Education Assessed by ACLS Checklist
Description: ACLS (Advanced Cardiac Life Support) score will be compared to score in first scenario to look for improvement. Items on the checklist were separated into two components: 1) the ACLS correct score (minimum score 0, maximum score 30), where higher scores indicate better performance, and 2) the ACLS risk score (minimum score 0, maximum score 17) where higher scores indicate worse performance. The mean difference in ACLS score between pre-test (scenario 1) and immediate post-test (scenario 2) is reported.
Time Frame: After managing second simulation scenario - Day 1
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | CRM Simulation
Number analyzed (Participants) | 48
Score on a scale
  ACLS correct score | 1.69 [0.78 to 2.56]
  ACLS risk score | -1.09 [-1.54 to -0.64]

5. Other Pre Specified Outcome: Retention of Learning From Simulation as Assessed by Ottawa Global Rating Scale
Description: Ottawa GRS score will be compared to score in second scenario on Day 1 to look for improvement. The Ottawa GRS assesses non-technical CRM skills on a 7-point scale (minimum 1, maximum 7), with higher scores indicating better performance. The mean difference in GRS score between immediate post-test (scenario 2) and retention post-test (scenario 3) is reported.
Time Frame: 3 months after completing first two scenarios - Day 90
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | CRM Simulation
Number analyzed (Participants) | 48
Score on a scale | -0.38 [-1.45 to 0.69]

6. Other Pre Specified Outcome: Retention of Learning From Simulation as Assessed by ACLS Checklist
Description: ACLS (Advanced Cardiac Life Support) score will be compared to score in second scenario on Day 1 to look for improvement. Items on the checklist were separated into two components: 1) the ACLS correct score (minimum score 0, maximum score 30), where higher scores indicate better performance, and 2) the ACLS risk score (minimum score 0, maximum score 17) where higher scores indicate worse performance. The mean difference in ACLS score between immediate post-test (scenario 2) and retention post-test (scenario 3) is reported.
Time Frame: 3 months after completing first two scenarios - Day 90
Measure: Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | CRM Simulation
Number analyzed (Participants) | 48
Score on a scale
  ACLS correct score | -0.34 [-1.31 to 0.64]
  ACLS risk score | 0.30 [-0.06 to 0.67]

ADVERSE EVENTS:
Time Frame: Three months.
Arm/Group | CRM Simulation
All-Cause Mortality (participants affected / at risk) | 0/48
Serious Adverse Events (participants affected / at risk) | 0/48
Other Adverse Events (participants affected / at risk) | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-19): https://cdn.clinicaltrials.gov/large-docs/47/NCT02683447/Prot_SAP_000.pdf